CLINICAL TRIAL: NCT00641329
Title: Phase III Evaluation of the Safety and Efficacy of CLONICEL (Clonidine HCl Sustained Release) as Add-on to Psychostimulant Medication vs. Psychostimulant Medication Alone in Children and Adolescents With ADHD
Brief Title: CLONICEL (Clonidine Sustained Release) as Add-on to Stimulant Medication in 6 to 17 Yr-olds With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addrenex Pharmaceuticals, Inc. (Industry)
Responsible Party: Moise Khayrallah, PhD / President & CEO, Addrenex Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLON-302
Record Dates: First submitted 2008-03-19; First posted 2008-03-24 (Estimated); Last update posted 2010-04-09 (Estimated); Status verified 2009-03

CONDITIONS: ADHD
Keywords: ADHD; ADD; Attention Deficit Hyperactivity Disorder; Attention Deficit; Clonidine; CLONICEL; Addrenex
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: CLONICEL (clonidine HCl sustained release)
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CLONICEL (clonidine HCl sustained release) — Flexible Dose (0.1 - 0.4 mg)
  Arms: 1
Drug: Placebo — Matching placebo tablets
  Arms: 2

SUMMARY:
The purpose of this study is to determine if CLONICEL (clonidine HCl sustained release) is a safe and effective add-on to psychostimulant therapy in children and adolescents with attention deficit hyperactivity disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Age 6-17 years, inclusive
* Diagnosis of ADHD
* Currently on a stable psychostimulant regimen for ADHD
* Lack of adequate response to stable psychostimulant regimen
* Ability to swallow tablets

Exclusion Criteria:

* Clinically significant illnesses or abnormalities upon evaluation
* Conduct Disorder
* Intolerance to clonidine
* History of seizures or syncope

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 198 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
ADHDRS-IV Total Score | Week 5
Treatment Emergent Adverse Events, Laboratory Tests, Vital Signs, and ECGs | Throughout Treatment and Follow-up Period

CONTACTS AND LOCATIONS:
Overall Officials: Moise Khayrallah, PhD, Study Director — Addrenex Pharmaceuticals
Locations (21):
- United States (21):
  - Little Rock, Arkansas
  - El Centro, California
  - Irvine, California
  - San Diego, California
  - Bradenton, Florida
  - Lauderhill, Florida
  - Miami, Florida
  - Bardstown, Kentucky
  - Baltimore, Maryland
  - St Louis, Missouri
  - Clementon, New Jersey
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Cleveland, Ohio
  - Oklahoma City, Oklahoma
  - Houston, Texas
  - Lake Jackson, Texas
  - Wharton, Texas
  - Clinton, Utah
  - Kirkland, Washington
  - Spokane, Washington